CLINICAL TRIAL: NCT02118584
Title: An Open-Label Extension and Safety Monitoring Study of Moderate to Severe Ulcerative Colitis Patients Previously Enrolled in Etrolizumab Phase II/III Studies
Brief Title: Study for Participants With Ulcerative Colitis Previously Enrolled in Etrolizumab Phase II/III Studies
Acronym: COTTONWOOD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to program discontinuation, based on mixed efficacy results in the parent studies. There were no safety concerns.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA28951; 2013-004435-72 (EudraCT Number)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1: Open-label Extension (Experimental): Participants with moderate to severe UC who were enrolled in the Phase II OLE study or the Phase III studies, and who meet the eligibility criteria for enrollment will receive open-label etrolizumab in Part 1 (OLE).
  Interventions: Drug: Etrolizumab
- Part 2: Safety Monitoring (No Intervention): All participants from Part 1 (OLE), participants whose PML follow-up is not completed within the Phase II OLE study, and participants transferring from the Phase III double-blind studies after the 12-week safety follow-up will be monitored for PML (92 weeks).

INTERVENTIONS:
Drug: Etrolizumab — Participants will receive etrolizumab 105 milligrams (mg), administered subcutaneously (SC) every 4 weeks for up to 9 years or until either commercial availability or the Sponsor's decision to terminate the study.
  Other Names: RG7413; RO5490261; PRO145223; rhuMAb Beta7
  Arms: Part 1: Open-label Extension

SUMMARY:
This two-part, part 1: open-label extension (OLE) and part 2: safety monitoring (SM) study will examine the efficacy and safety of continued etrolizumab treatment in moderate to severe ulcerative colitis (UC) participants previously enrolled in etrolizumab Phase II/III studies. Participants with moderate to severe UC who were enrolled in the Phase II OLE study (GA27927 [NCT01461317]) or the Phase III studies (GA28948 [NCT02163759], GA28949 [NCT02171429], GA28950 [NCT02100696], GA29102 [NCT02165215], and GA29103 [NCT02136069]) were included. Participants from the Phase II OLE study or the Phase III studies who are not eligible or willing to receive etrolizumab in the OLE-SM study, and who have completed the 12-week safety follow-up period will be enrolled in Part 2. Part 1 of OLE-SM will continue for up to 9 years after the first participant is enrolled into the study. Following Part 1, participants will enter Part 2 for a period of 92 weeks.

ELIGIBILITY:
Inclusion Criteria:

Part 1 (Open-label Extension)

- Participants previously enrolled in the Phase II OLE study or Phase III controlled studies who meet the eligibility criteria for open-label etrolizumab for those studies as described in the protocol

Part 2 (Safety Monitoring)

* Participants whose safety follow-up or PML follow-up is not completed within Study GA27927 and participants who had their last dose of etrolizumab in July 2016 in Study GA27927 and are not eligible or willing to enroll in Part 1 (OLE)
* Participants who participated in one of the etrolizumab Phase III studies and are not eligible or willing to enter Part 1 (OLE)
* Participants who transfer from Part 1 (OLE)
* Completion of the 12-week safety follow-up prior to entering.

Exclusion Criteria:

Part 1 (Open-label Extension)

* Withdrawal of consent from and participant not compliant in the Phase II OLE study or any of the Phase III studies
* Participant who discontinued etrolizumab/etrolizumab placebo prior to Week 10 or did not perform the Week 10 visit of the Phase III Studies GA28948, GA28949, GA29102, and GA29103
* Participant who discontinued etrolizumab/etrolizumab placebo prior to Week 14 or did not perform the Week 14 visit of the Phase III Study GA28950
* Any new, significant, uncontrolled condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1822 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (411):
- United States (57):
  - University of Alabama Medical Center, Birmingham, Alabama
  - University of California San Diego Medical Center, La Jolla, California
  - University of California, Irvine Medical Center, Orange, California
  - SDG Clinical Research, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Ventura Clinical Trials, Ventura, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Rocky Mountain Gastroenterology Associates, Wheat Ridge, Colorado
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Regenerate Clinical Trials, Miami, Florida
  - IMIC, Inc, Miami Beach, Florida
  - FQL Research, LLC, Miramar, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - University of Chicago Medical Center; Medicine, Section of Pulmonary, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Aquiant Research, New Albany, Indiana
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Massachusetts General Hospital; Crohn's & Colitis Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Kansas City Research Institute, LLC, Kansas City, Missouri
  - Clinica Peruano Americana S.A., Great Neck, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical College (WCMC) - Judith Jaffe Multiple Sclerosis Center (JJMSC), New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Consultants for Clin. Rsrch, Cincinnati, Ohio
  - UC Health Clinical Trials Office; Division of Digestive Diseases, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastroenterology Center of the Midsouth, P.C., Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Wellness Clinical Research Center, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Ericksen Research and Development, Clinton, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - McGuire Research Institute; Gastroenterology, Richmond, Virginia
  - Washington Gastroenterology, Bellevue, Washington
- Argentina (2):
  - Instituto Medico DAMIC, Córdoba
  - Hospital Provincial del Centenario, Rosario
- Australia (14):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, Mackay, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Launceston General Hospital; Gastroenterology Research, Launceston, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
  - Royal Melbourne Hospital; Department of Colorectal Medicine and Genetics, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (9):
  - GZA Ziekenhuizen - Campus Sint-Vincentius, Antwerp
  - Imeldaziekenhuis, Bonheiden
  - CHU St Pierre (St Pierre), Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc; Pharmacy, Brussels
  - UZ Gent, Ghent
  - AZ Sint Elisabeth Herentals, Herentals
  - UZ Leuven; Neurology, Leuven
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (17):
  - Hospital Universitario Walter Cantidio - UFC, Fortaleza, Ceará
  - Hospital Universitario Prof Edgar Santos-Ufba; Ambulatorio Magalhaes Neto 3Andar- Dermatologia, Salvador, Estado de Bahia
  - CCBR - Brasilia, Brasília, Federal District
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital Universitario Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - CAEP - Centro Avancado de Estudos e Pesquisas Ltda., Campinas, São Paulo
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Pesquisare Saúde Sociedade Simples, Santo André, São Paulo
  - Hospital Estadual Mario Covas, São Bernardo do Campo, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual/HSPE-SP, São Paulo, São Paulo
- Bulgaria (12):
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - DCC Sv. Pantaleymon OOD; II-nd Clinic of Neurology, Pleven
  - Medical center Medconsult Pleven OOD, Pleven
  - MHAT - Ruse, AD, Rousse
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - "City Clinic UMHAC" EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL, EAD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - MHAT 'Sv. Marina', EAD; First Children's Clinic, Varna
  - MC Medica Plus, Veliko Tarnovo
- Canada (14):
  - University of Calgary, Calgary, Alberta
  - Zeidler Ledcor Centre - University of Alberta; Division of Gasroenterology, Edmonton, Alberta
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Gastroenterology Research, Halifax, Nova Scotia
  - Guelph GI & Surgery Clinic, Guelph, Ontario
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - Centre de santé et de services sociaux Champlain-Charles-Le Moyne, Greenfield Park, Quebec
  - Hotel Dieu de Levis, Lévis, Quebec
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Colombia (2):
  - RTS - Fundación Valle de Lili, Cali
  - Instituto de Coloproctologia ICO S.A.S., Medellín
- Croatia (2):
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Sveti Duh; Department of Neurology, Zagreb
- Czechia (12):
  - Vojenska nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne; I.Interni kardioangiologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Oblastni nemocnice Kladno, a.s., nemocnice Stredoces. kraje; Endoskopicke centrum, Kladno
  - PreventaMed, s.r.o., Olomouc
  - Mestska Nemocnice Ostrava, Ostrava
  - Pardubicka krajska nemocnice a.s., Pardubice
  - ISCARE a.s., Prague
  - Nemocnice Na Bulovce, Prague
  - Krajska zdravotni, a.s. ? Masarykova nemocnice v Usti nad Labem, o.z., Ocni oddeleni, Ústí nad Labem
  - Krajska nemocnice T. Bati, a.s., Zlín
- Denmark (3):
  - Ålborg Universitets Hospital; Gastromedicinsk, Aalborg
  - Herlev og Gentofte Hospital, Hellerup
  - Rigshospitalet; Afdeling for Tarmsvigt og Leversygdomme, København Ø
- Estonia (5):
  - OÜ Innomedica, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (14):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU de Caen Hopital Cote de Nacre, Caen
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Hôpital Beaujon, Clichy
  - Hopital Claude Huriez - CHU Lille, Lille
  - CHU Hopital Saint Eloi, Montpellier
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hôpital Saint-Louis, Paris
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud; Service de Gastro-Enterologie, Pierre-Bénite
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Höpital Hautepierre; Pediatrie1, Strasbourg
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (20):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil GmbH, Bochum
  - Universitaetsklinikum Erlangen, Erlangen
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg; Urology, Freiburg im Breisgau
  - Universitaetsklinikum Halle (Saale), Halle
  - Hamburgisches Forschungsinstitut fuer CED, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Gastroenterologie Eppendorfer Baum, Hamburg
  - Medizinische Hochschule Hannover; Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitaetsklinikum Jena; Apotheke des Uniersitätsklinikums Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Medizinisches Zentrum Klinikum Lueneburg, Lüneburg
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Universitaetsklinikum Muenster, Münster
  - Gemeinschaftspraxis Dres. Joachim Mueller und Steffi Appelt, Schweinfurt
  - Universitaetsklinikum Ulm, Ulm
- University General Hospital of Heraklion, Heraklio, Greece
- University of Hong Kong, Hong Kong, Hong Kong
- Hungary (16):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba
  - Semmelweis Egyetem; Belgyogyaszati es Hematologiai Klinika, Budapest
  - Eszak-Kozep-budai Centrum, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Pannónia Klinika Magánorvosi, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont; Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest
  - Endomedix Diagnosztikai Kozpont, Budapest
  - Vasutegeszsegugyi Kft. - Debreceni Egeszsegugyi Kozpont, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Markhot Ferenc Oktato Korhaz es Rendelointezet, Eger
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Pecsi Tudomanyegyetem, Pécs
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- India (10):
  - Deccan College of Medical Sciences and Allied Hospitals; Department of Gastroenterology, Hyderabad, Andhra Pradesh
  - Nirmal Hospital, Surat, Gujarat
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - M. S. Ramaiah Medical College and Hospital, Bengaluru, Karnataka
  - Kasturba Medical College & Hospital, Manglore, Karnataka
  - Midas institute of Gastroenterology, Nagpur, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - S. R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - King Edward Memorial Hospital Research Centre, Pune
- Israel (8):
  - Bnai Zion Medical Center; Internal Medicine, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center Beilinson Campus; Gaucher Clinic Genetics Institute, Petach Tiqwa
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh, Rishon LeZiyyon
  - Chaim Sheba Medical Center; Pediatrics B North and Pediatric Endocrinology Unit, Tel Litwinsky
- Italy (19):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpigh, Bologna, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Ospedale Sandro Pertini, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Lombardy
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan, Lombardy
  - Ospedale di Circolo; Neuropsichiatria Infantile, Rho, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Lombardy
  - IRCCS Ospedale Casa Sollievo della Soffenza; Stru Comp di Gastroenterologia ed Endoscopia digest, San Giovanni Rotondo, Lombardy
  - Ospedale Mauriziano Umberto I, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Latvia (3):
  - Central Outpatient Clinic, Daugavpils
  - Pauls Stradins Clinical University Hospital, R?ga
  - Digestive Diseases Center "Gastro", R?ga
- Lithuania (3):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Klaipeda Seamen's Hospital, Public Institution, Klaipėda
  - Vilnius University Hospital Santariskiu Clinic, Public Institution; Cardiology, Vilnius
- Malaysia (4):
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - University Malaya Medical Center, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Perempuan Zainab II; Department of Medicine, Kota Bharu
- Mexico (5):
  - Centro Integral en Reumatología S.A. de C.V. (CIRSA), Guadalajara, Jalisco
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Hospital Universitario Dr Jose Eleuterio Gonzalez; Universidad Autónoma de Nuevo León, Monterrey, Nuevo León
  - Centro Regiomontano de Estudios Clínicos Roma S.C., Monterrey, Nuevo León
  - Phylasis Clinicas Research S de RL de CV, Cuautitlán Izcalli
- Netherlands (3):
  - Amsterdam UMC Location VUMC, Amsterdam
  - Amsterdam UMC Location AMC, Amsterdam
  - Radboudumc, NL -nijmegen
- New Zealand (6):
  - North Shore Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Shakespeare Specialist Group, Takapuna
  - Tauranga Hospital, Tauranga
- Akershus universitetssykehus HF, Lørenskog, Norway
- Poland (28):
  - AppleTreeClinics Sp. z o.o., ?ód?
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka, Chojnice
  - Centrum Medyczne Sw. Lukasza, Cz?stochowa
  - 7 Szpital Marynarki Wojennej z Przychodnia SPZOZ im. W. Lasinskiego, Gdansk
  - Pro Familia Altera Sp z o.o., Katowice
  - Nzoz All-Medicus, Katowice
  - Uniwersyteckie Centrum Kliniczne im. prof. K. Gibinskiego SUM, Katowice
  - NZOZ Centrum Medyczne ProMiMed, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med, Ksawerów
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lublin
  - GASTROMED Sp. z o.o., Lublin
  - Allmedica Badania Kliniczne Sp z o.o. Sp K., Nowy Targ
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - SOLUMED Centrum Medyczne, Późna
  - Centrum Medyczne Medyk, Rzeszów
  - Gabinet Lekarski, Bartosz Korczowski, Rzeszów
  - Specjalistyczna Praktyka Lekarska Dr med. Marek Horynski; endoskopia, Sopot
  - Niepubliczny Zaklad Opieki Zdrowotnej SONOMED, Szczecin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Zespó Przychodni Specjalistycznych PRIMA, Warsaw
  - Endoterapia PFG Sp. z o.o., Warsaw
  - Narodowy Instytut Onkologii im. Marii Sk?odowskiej-Curie - Pa?stwowy Instytut Badawczy, Warsaw
  - Nzoz Vivamed, Warsaw
  - Przychodnia EuroMediCare, Wroc?aw
  - PlanetMed, Wroc?aw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Portugal (2):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
- Romania (4):
  - S.C MedLife S.A, Bucharest
  - Centrul Medical Unirea SRL, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (23):
  - Yusupov Hospital, Moskva, Adygeya Republic
  - SBEI HPE Altai StateMedicalUniversityofMoH andSD, Barnaul, Altayskiy Kray
  - FSBIH Central Clinical Hospital of RAS, Moscow, Moscow Oblast
  - FSBI ?State Scientific Centre of Coloproctology" of the MoH of RF; Gastroenterology, Moscow, Moscow Oblast
  - SBHI of NN region ?RCH of NN n.a. N.A.Semashko?, Nizhny Novgorod, Niznij Novgorod
  - SEIHPE "Rostov SMU of MoH of RF", Rostov-on-Don, Rostov Oblast
  - FSBMEI HPE "Military Medical Academy n.a. S.M. Kirov" of the MoD of the RF; Therapy, Saint Petersburg, Sankt-Peterburg
  - FFSBI "The Nikiforov Russian Center of Emergency and Radiation Medicine"; Pulmonology, Saint Petersburg, Sankt-Peterburg
  - SPb SBIH "City Multy-field Hospital # 2"; Intensive Pulmonology and Thoracal Surgery, Saint Petersburg, Sankt-Peterburg
  - Baltic Medicine, Saint Petersburg, Sankt-Peterburg
  - City Hospital #26, Saint Petersburg, Sankt-Peterburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg, Sankt-Peterburg
  - SBIH City Clinical Hospital #31, Saint Petersburg, Sankt-Peterburg
  - SPb SHI "City Hospital #9", Saint Petersburg, Sankt-Peterburg
  - LLC International Medical Centre ?SOGAZ?, Saint Petersburg, Sankt-Peterburg
  - Medical and Sanitary Division of Severstal, Cherepovets, Vologda Oblast
  - SBEI HPE "Voronezh State Medical University n.a. N.N. Burdenko" of the MoH of the RF, Voronezh, Voronez
  - Irkutsk State Medical Academy of Continuing Education, Irkutsk
  - FSBI "Scientific Research Institute of Physyology and Basic Medicine" under the SB of RAMS, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - SBEI of HPE "Omsk SMA" Ministry of healthcare of RF", Omsk
  - Stavropol Regional Clinical Diagnostic Consultative Center, Stavropol
  - FSBEI HE "Stavropol State Medical University" of Ministry of Healthcare of Russian Federation, Stavropol
- Serbia (5):
  - Clinical Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Djordje Joanovic, Zrenjanin
- Singapore General Hospital, Singapore, Singapore
- Slovakia (7):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Nemocnica A.Lena Humenne, n.o., Humenné
  - Endomed, s.r.o., Košice
  - KM Management spol. s r.o., Nitra
  - Gastro I, s.r.o., Prešov
  - Svet zdravia a.s., Rimavská Sobota
  - Accout Center s.r.o., Šahy
- South Africa (4):
  - Netcare Universitas Private Hospital, Bloemfontein
  - Dr MJ Prins Practice, Cape Town
  - Dr JP Wright Practice, Cape Town
  - Emmed Research, Pretoria
- South Korea (17):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam Univ. Hospital, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - CHA Bundang Medical Centre; CHA university, Seongnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center., Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Fundacion Hospital de Alcorcon; Servicio de Digestivo, Alcorcón, Madrid
  - Centro Médico Teknon, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (2):
  - Inselspital-Universitaetsspital Bern, Bern
  - Crohn-Colitis Zentrum Bern - Gemeinschaftspraxis Balsiger, Seibold und Partner, Bern
- Turkey (Türkiye) (3):
  - Gazi University Medical Faculty; Gastroenterology, Ankara
  - Haydarpasa Numune Training and Research Hospital; Medical Oncology, Istanbul
  - Kocaeli Universitesi Tip Fakultesi; Infectious Diseases, Kocaeli
- Ukraine (29):
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv, Kharkiv Governorate
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv, Kharkiv Governorate
  - Communal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv, Kharkiv Governorate
  - CI of SRC Sumy RCH Dept of Gasroenterology Sumy SU MI, Sumy, Kharkiv Governorate
  - LLC Gastroenterology Center IBD Team, Zaporizhzhia, Kharkiv Governorate
  - CNE Kyiv CCH #18, Kyiv, KIEV Governorate
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv, KIEV Governorate
  - Medical Center of Limited Liability Company Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - Med Center of International Institute of Clinical Trials LLC; Medical Center "OK!Clinic+", Kyiv, KIEV Governorate
  - CI of Kyiv RC Regional Clinical Hospital #2, Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital, Lviv, KIEV Governorate
  - CI UDH Dept of Ther SHEI Fac of PGE&Pre-Univ Training, Uzhhorod, KIEV Governorate
  - A.Novak Transcarpathian Regional Clinical Hospital, Uzhhorod, KIEV Governorate
  - RCNECRCH Dept of Surgery, SHEI Ukr BSMU, Chernivtsi, Podolia Governorate
  - CI City Hospital #1, Zaporizhzhia, Tavria Okruha
  - RCI Chernivtsi RCH Gastroenterology Bukovinsky SMU, Chernivtsi
  - SI Dnipropetrovsk MA of MOHU SI Institute of gastroenterology of AMSU, Dnipropetrovsk
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - CI of Healthcare Kharkiv CCH #13, Kharkiv
  - CI Kherson Afanasii and Olha Tropiny City Clinical Hospital, Kherson
  - CNI Consultative and Diagnostic Center of Desnianskyi District of Kyiv, Kyiv
  - Odessa regional clinical Hospital, Odesa
  - M.V. Sklifosovskyi Poltava RCH Dept of Gastroenterology HSEIU UMSA, Poltava
  - M.V. Sklifosovskyi Poltava RCH Outpatient UMSA HSEIU Ukrainian Medical Stomatological Academy, Poltava
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - MCIC Health Clinic BO LTD TPC Slaomed, Vinnytsia
  - Co Ltd. Diaservice, Zaporizhzhia
  - CI City Hospital #7, Zaporizhzhia
- United Kingdom (12):
  - Addenbrooke's Hospital, Cambridge
  - University Hospital Coventry, Coventry
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - St James University Hospital, Leeds
  - The Royal London Hospital, London
  - University College London Hospital, London
  - St Thomas Hospital, London
  - King's College London, London
  - Fairfield General Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals; QMC Campus, Nottingham
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study in 42 countries. All participants who were enrolled in this study previously took part in one of the following parent studies - Phase II: GA27927; Phase III: GA28948, GA28949, GA28950, GA29102, GA29103.
Pre-assignment Details: This study consists of two parts, Part 1: Open-label extension (OLE) period and Part 2: Progressive multifocal leukoencephalopathy (PML) safety monitoring (SM) period. A total of 1822 participants with ulcerative colitis (UC) were enrolled in the study, 1773 participants in Part 1 and 796 participants in Part 2. Of the 796, 49 participants were directly enrolled into the Part 2: PML SM period from their respective parent studies.
Groups:
- Part 1 (OLE): Etrolizumab Only: Participants received etrolizumab 105 milligrams (mg), subcutaneously (SC) every 4 weeks (Q4W) for maximum of 369.9 weeks, followed by a 12-week safety follow-up.
- Part 1 (OLE) to Part 2 (PML SM): Participants received etrolizumab 105 mg, SC, Q4W for maximum of 369.9 weeks, followed by a 12-week safety follow-up in the OLE period. After the OLE period, participants were given the option to enter Part 2 (PML SM). Participants who chose to enter the PML SM period were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
- Part 2 (PML SM) Only: Participants from the Phase II or Phase III studies who were not eligible/did not wish to enroll in Part 1 (OLE), and had completed the 12-week safety follow-up period in their parent study were enrolled directly in Part 2 (PML SM). Participants were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
Period: Part 1: Open Label Extension Period
Arm/Group | Part 1 (OLE): Etrolizumab Only | Part 1 (OLE) to Part 2 (PML SM) | Part 2 (PML SM) Only
Started | 1026 | 747 | 0
Completed | 9 | 747 | 0
Not Completed | 1017 | 0 | 0
Not completed — Adverse Event | 79 | 0 | 0
Not completed — Death | 9 | 0 | 0
Not completed — Lost to Follow-up | 53 | 0 | 0
Not completed — Non-compliance | 12 | 0 | 0
Not completed — Other | 135 | 0 | 0
Not completed — Physician Decision | 128 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 29 | 0 | 0
Not completed — Other | 3 | 0 | 0
Not completed — Withdrawal by Subject | 568 | 0 | 0
Period: Part 2: PML Safety Monitoring Period
Arm/Group | Part 1 (OLE): Etrolizumab Only | Part 1 (OLE) to Part 2 (PML SM) | Part 2 (PML SM) Only
Started | 0 | 747 | 49
Completed | 0 | 317 | 43
Not Completed | 0 | 430 | 6
Not completed — Adverse Event | 0 | 5 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 22 | 3
Not completed — Non-Compliance | 0 | 0 | 1
Not completed — Reason Not Specified | 0 | 6 | 0
Not completed — Physician Decision | 0 | 10 | 1
Not completed — Study Terminated by Sponsor | 0 | 354 | 0
Not completed — Withdrawal by Subject | 0 | 32 | 1

BASELINE CHARACTERISTICS:
Population: All Patients Population included all participants who were enrolled in the study.
Groups:
- Part 1 (OLE): Etrolizumab Only: Participants received etrolizumab 105 mg, SC, Q4W for maximum of 369.9 weeks, followed by a 12-week safety follow-up.
- Total: Total of all reporting groups
Arm/Group | Part 1 (OLE): Etrolizumab Only | Part 1 (OLE) to Part 2 (PML SM) | Part 2 (PML SM) Only | Total
Number analyzed (Participants) | 1026 | 747 | 49 | 1822
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (13.3) | 40.7 (14.1) | 42.7 (15.2) | 40.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 417 | 333 | 23 | 773
  Male | 609 | 414 | 26 | 1049
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 93 | 0 | 152
  Not Hispanic or Latino | 915 | 632 | 47 | 1594
  Unknown or Not Reported | 52 | 22 | 2 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 101 | 40 | 4 | 145
  Black or African American | 11 | 18 | 0 | 29
  White | 843 | 635 | 40 | 1518
  Other | 36 | 32 | 2 | 70
  Multiple | 1 | 1 | 0 | 2
  Unknown | 33 | 20 | 2 | 55

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Clinical Remission as Determined by the Partial Mayo Clinic Score (pMCS)
Description: The pMCS is a composite of 3 assessments, each rated from 0 (none) to 3 (severe disease): stool frequency, rectal bleeding, and physician's global assessment. The total score for pMCS ranges from 0 (none) to 9 (severe disease). pMCS clinical remission was defined as pMCS ≤ 2, a rectal bleeding score of 0-1, physician's global assessment of 0-1, stool frequency subscore of 0-1. Percentages have been rounded off.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, 204, 216, 228, 240, 252, 264, 276, 288, 300, 312 and 324 weeks
Population: OLE Population included all participants who received at least one dose of open label etrolizumab in Part 1 of the study. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Number; unit: percentage of participants
Groups:
- Part 1 (OLE): Etrolizumab: Participants received etrolizumab 105 mg, SC, Q4W for maximum of 369.9 weeks, followed by a 12-week safety follow-up.
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1772
percentage of participants
  Baseline | 32.0
  Week 4: number analyzed (Participants) | 1365
  Week 4 | 47.2
  Week 8: number analyzed (Participants) | 1302
  Week 8 | 52.2
  Week 12: number analyzed (Participants) | 1292
  Week 12 | 55.9
  Week 24: number analyzed (Participants) | 935
  Week 24 | 63.7
  Week 36: number analyzed (Participants) | 879
  Week 36 | 68.3
  Week 48: number analyzed (Participants) | 856
  Week 48 | 73.4
  Week 60: number analyzed (Participants) | 810
  Week 60 | 72.2
  Week 72: number analyzed (Participants) | 768
  Week 72 | 75.4
  Week 84: number analyzed (Participants) | 733
  Week 84 | 76.5
  Week 96: number analyzed (Participants) | 718
  Week 96 | 77.2
  Week 108: number analyzed (Participants) | 665
  Week 108 | 72.0
  Week 120: number analyzed (Participants) | 593
  Week 120 | 77.4
  Week 132: number analyzed (Participants) | 535
  Week 132 | 82.2
  Week 144: number analyzed (Participants) | 501
  Week 144 | 80.0
  Week 156: number analyzed (Participants) | 461
  Week 156 | 78.5
  Week 168: number analyzed (Participants) | 410
  Week 168 | 81.0
  Week 180: number analyzed (Participants) | 378
  Week 180 | 78.8
  Week 192: number analyzed (Participants) | 355
  Week 192 | 80.8
  Week 204: number analyzed (Participants) | 318
  Week 204 | 83.6
  Week 216: number analyzed (Participants) | 289
  Week 216 | 84.8
  Week 228: number analyzed (Participants) | 262
  Week 228 | 85.1
  Week 240: number analyzed (Participants) | 230
  Week 240 | 82.6
  Week 252: number analyzed (Participants) | 207
  Week 252 | 86.0
  Week 264: number analyzed (Participants) | 164
  Week 264 | 84.8
  Week 276: number analyzed (Participants) | 150
  Week 276 | 86.0
  Week 288: number analyzed (Participants) | 136
  Week 288 | 82.4
  Week 300: number analyzed (Participants) | 90
  Week 300 | 86.7
  Week 312: number analyzed (Participants) | 62
  Week 312 | 87.1
  Week 324: number analyzed (Participants) | 30
  Week 324 | 80.0

2. Primary Outcome: Part 1: Percentage of Participants With Remission as Determined by the Mayo Clinic Score (MCS)
Description: The Mayo Clinic scoring system is a composite of 4 assessments for UC disease activity. The 4 component sub-scores are: 1) stool frequency, 2) rectal bleeding, 3) flexible sigmoidoscopy scores, and 4) physician's global assessment, each rated from 0-3, 0 representing no pathology to 3 for severe disease. The minimum Mayo Score is 0 (no pathology) and the maximum is 12 (severe disease). MCS remission was defined as MCS ≤ 2, a rectal bleeding score of 0, physician's global assessment of 0-1, stool frequency subscore of 0-1 and endoscopy score of 0-1. Percentage has been rounded off.
Time Frame: At OLE Week 108
Population: OLE Population included all participants who received at least one dose of open label etrolizumab in Part 1 of the study. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 623
percentage of participants | 58.1

3. Primary Outcome: Part 1: Percentage of Participants With Endoscopic Remission
Description: The Mayo scoring system is a composite of 4 assessments for UC disease activity. The 4 component sub-scores are: 1) stool frequency, 2) rectal bleeding, 3) flexible sigmoidoscopy scores, and 4) physician's global assessment, each rated from 0-3, 0 representing no pathology to 3 for severe disease. The minimum Mayo Score is 0 (no pathology) and the maximum is 12 (severe disease). Endoscopic remission was defined as Mayo Endoscopic subscore = 0. Percentage has been rounded off.
Time Frame: At OLE Week 108
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 900
percentage of participants | 45.7

4. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Severity of AEs Assessed Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 [NCI CTCAE v4.0]
Description: An AE is any untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. AEs were graded as per NCI CTCAE v4.0. Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4=Life-threatening consequences/urgent intervention indicated; Grade 5=Death related to adverse event.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: OLE Population included all participants who received at least one dose of open label etrolizumab in Part 1 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants
  Any AEs | 1431
  Grade 1 AEs | 315
  Grade 2 AEs | 679
  Grade 3 AEs | 405
  Grade 4 AEs | 23
  Grade 5 AEs | 9

5. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigation, whether or not considered related to the medicinal (investigational) product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants | 373

6. Primary Outcome: Part 1: Number of Participants With Infection Related AEs and Severity of Infection-Related AEs Assessed Using NCI CTCAE v4.0
Description: An AE is any untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. AEs were graded as per NCI CTCAE v4.0. Grade 1= Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living; Grade 4=Life-threatening consequences/urgent intervention indicated; Grade 5=Death related to adverse event.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants
  Infection Related AEs, Any Grade | 825
  Infection Related AEs, Grade 1 | 576
  Infection Related AEs, Grade 2 | 423
  Infection Related AEs, Grade 3 | 96
  Infection Related AEs, Grade 4 | 6
  Infection Related AEs, Grade 5 | 1

7. Primary Outcome: Part 1: Number of Participants With Serious Infection Related AES
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants | 110

8. Primary Outcome: Part 1: Number of Participants With Injection Site Reactions and Severity of Injection Site Reactions Assessed Using NCI CTCAE v4.0
Description: AE=untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. Injection-site reaction=any local reaction occurring at the site of injection following study drug administration. Signs (e.g., erythema, induration/swelling at injection site) and symptoms (e.g., pain, pruritus at injection site). Injection site reactions. were graded as per NCI CTCAE v4.0. Grade 1=Tenderness with or without associated symptoms (e.g., warmth, erythema, itching); Grade 2=Pain; lipodystrophy; edema; phlebitis; Grade 3=Ulceration or necrosis; severe tissue damage; operative intervention indicated; Grade 4=life-threatening consequences or urgent intervention indicated; Grade=5 death related to AE.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants
  Injection Site Reactions, Any Grade | 32
  Injection Site Reactions, Grade 1 | 28
  Injection Site Reactions, Grade 2 | 5
  Injection Site Reactions, Grade 3 | 0
  Injection Site Reactions, Grade 4 | 0
  Injection Site Reactions, Grade 5 | 0

9. Primary Outcome: Part 1: Number of Participants With AEs Leading to Etrolizumab Discontinuation
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a Etrolizumab, whether or not considered related to the medicinal (investigational) product. Number of participants who discontinued etrolizumab treatment during the OLE period have been reported here.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants | 234

10. Primary Outcome: Part 1: Number of Participants With Malignancies
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. Number of participants who developed malignancies during the OLE period have been reported here.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants | 38

11. Primary Outcome: Part 1: Number of Participants With Hypersensitivity Reactions and Severity of Hypersensitivity Assessed Using NCI-CTCAE v4.0
Description: AE=untoward medical occurrence in participant administered a pharmaceutical product & regardless of causal relationship with this treatment. AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. Hypersensitivity was assessed as per NCI CTCAE v4.0. Grade 1=Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated; Grade 2=Moderate; minimal, local or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living; Grade 3=Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living.
Time Frame: From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (OLE): Etrolizumab
Number analyzed (Participants) | 1773
Participants
  Hypersensitivity Reactions, Any Grade | 85
  Hypersensitivity Reactions, Grade 1 | 65
  Hypersensitivity Reactions, Grade 2 | 19
  Hypersensitivity Reactions, Grade 3 | 4

12. Primary Outcome: Part 2: Number of Participants With Confirmed Progressive Multifocal Leukoencephalopathy (PML) During the Post-Treatment PML Monitoring Period
Time Frame: From end of safety follow-up in Part 1 or Phase II/III parent studies up to a maximum of 92 weeks
Population: PML Safety Monitoring population included all participants who entered the PML SM period. No treatment was administered in PML SM period, and hence participants entering from Part 1 (OLE) and the parent studies have been reported together.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: PML-SM: Participants from Phase II or Phase III studies who were not eligible/did not wish to enroll in Part 1 (OLE), and had completed the 12-week safety follow-up period in their parent study were enrolled directly in Part 2 (PML SM). Participants were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
Arm/Group | Part 2: PML-SM
Number analyzed (Participants) | 796
Participants | 0

ADVERSE EVENTS:
Time Frame: Part 1 (OLE): From Day 1 up to end of 12-week safety follow up in OLE (approximately 7 years); Part 2 (PML SM): From end of safety follow-up in Part 1 or Phase II/III parent studies up to a maximum of 92 weeks
Description: OLE population included all participants who received at least one dose of open label etrolizumab in Part 1 of the study. PML SM population included all participants who entered the PML SM period. Part 2: PML SM arm includes all participants who entered PML SM from Part 1 (OLE) and from their respective parent studies. No treatment was administered in PML SM period, and hence participants entering from Part 1 (OLE) and the parent studies have been reported together.
Groups:
- Part 2 (PML SM): Participants from Part 1 (OLE) and from Phase II/III studies who were not eligible/did not wish to enroll in Part 1 (OLE) and had completed the 12-week safety follow-up period were enrolled in the Part 2 (PML SM). Participants were monitored for PML for a maximum of 92-weeks, during which no etrolizumab treatment was administered.
Arm/Group | Part 1 (OLE): Etrolizumab | Part 2 (PML SM)
All-Cause Mortality (participants affected / at risk) | 9/1773 | 1/796
Serious Adverse Events (participants affected / at risk) | 373/1773 | 2/796
Other Adverse Events (participants affected / at risk) | 1052/1773 | 2/796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (OLE): Etrolizumab (N=1773) | Part 2 (PML SM) (N=796)
Anaemia (Blood and lymphatic system disorders) | 16 (19) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tethered oral tissue (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 3 (3) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 131 (153) | 1 (1)
Colon dysplasia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malocclusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (3) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 7 (7) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 11 (11) | 0 (0)
Bacterial infection (Infections and infestations) | 2 (3) | 0 (0)
Bacterial salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 13 (13) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 0 (0)
Complicated appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Coronavirus infection (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (2) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 3 (4) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Focal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 3 (3) | 0 (0)
Latent tuberculosis (Infections and infestations) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Meningitis listeria (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Rectal abscess (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spondylolysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon laxity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papillary breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 10 (14) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 5 (6) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Paraphimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Granuloma skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (OLE): Etrolizumab (N=1773) | Part 2 (PML SM) (N=796)
Anaemia (Blood and lymphatic system disorders) | 128 (149) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 98 (117) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 587 (882) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 95 (114) | 0 (0)
COVID-19 (Infections and infestations) | 165 (178) | 0 (0)
Influenza (Infections and infestations) | 100 (121) | 0 (0)
Nasopharyngitis (Infections and infestations) | 226 (344) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 110 (157) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 128 (172) | 0 (0)
Headache (Nervous system disorders) | 134 (187) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT02118584/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT02118584/SAP_001.pdf